CLINICAL TRIAL: NCT01022775
Title: Assessment of Dynamic Humeral Centering in Impingement Syndrome: a Randomized Clinical Trial
Brief Title: Dynamic Humeral Centering in Impingement Syndrome
Acronym: ADHCIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Societe Francaise de Rhumatologie (Other)
Responsible Party: Thérèse NGOUE, Department of clinical research and development
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P000203; CRC99241 (Other: Department of clinical research and development)
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Degenerative Rotator Cuff Disease With Impingement Syndrome
Keywords: Degenerative rotator cuff disease; Impingement syndrome; Dynamic humeral centering; Randomized clinical trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Dynamic humeral centering (Experimental): Dynamic humeral centering performed for 6 weeks, in 15 supervised individual outpatient sessions, plus daily home exercises for 12 months.
  Interventions: Procedure: Dynamic humeral centering
- 2: Nonspecific mobilisation (Active Comparator): Nonspecific mobilisation performed for 6 weeks, in 15 supervised individual outpatient sessions, plus daily home exercises for 12 months.
  Interventions: Procedure: Nonspecific mobilisation

INTERVENTIONS:
Procedure: Dynamic humeral centering — Dynamic humeral centering performed for 6 weeks, in 15 supervised individual outpatient sessions, plus daily home exercises for 12 months.
  Arms: 1: Dynamic humeral centering
Procedure: Nonspecific mobilisation — Nonspecific mobilisation performed for 6 weeks, in 15 supervised individual outpatient sessions, plus daily home exercises for 12 months.
  Arms: 2: Nonspecific mobilisation

SUMMARY:
The purpose of this study is to determine wether dynamic humeral centering is effective in patients with impingement syndrome of the shoulder

DETAILED DESCRIPTION:
Clinical trial with randomization for treatment and physiotherapist

ELIGIBILITY:
Inclusion Criteria:

* age > 30 years
* pain duration > 1 month
* presence of at least 2 positive impingement test results from Neer, Yocum and Hawkins testing
* total Constant score < 80.

Exclusion Criteria: concerning the shoulder

* stiffness
* anteroposterior instability
* tendinous calcification
* corticosteroid injection within the previous 30 days
* previous surgery
* humeral fracture
* inflammatory joint disease
* neoplastic disorders

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2001-04; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Constant total score as a mean and by category | at 3 months

SECONDARY OUTCOMES:
Constant total score | at 12 months
Constant subscores for pain, activity, mobility and strength, and self-assessed disability on a 0- to 100-point visual analog scale, and analgesic and nonsteroidal anti-inflammatory drug (NSAID) use | at 3 months
Constant subscores for pain, activity, mobility and strength, and self-assessed disability on a 0- to 100-point visual analog scale, and analgesic and nonsteroidal anti-inflammatory drug (NSAID) use | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Johann BEAUDREUIL, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Rheumatology, Lariboisière Hospital, Paris, France

REFERENCES:
- [Derived] Beaudreuil J, Ostertag A, Lasbleiz S, Vicaut E, Yelnik A, Bardin T, Orcel P. Efficacy of dynamic humeral centering according to Neer test results: a stratified analysis of a randomized-controlled trial. Int J Rehabil Res. 2015 Mar;38(1):81-3. doi: 10.1097/MRR.0000000000000079. PMID 25185788
- [Derived] Beaudreuil J, Lasbleiz S, Richette P, Seguin G, Rastel C, Aout M, Vicaut E, Cohen-Solal M, Liote F, de Vernejoul MC, Bardin T, Orcel P. Assessment of dynamic humeral centering in shoulder pain with impingement syndrome: a randomised clinical trial. Ann Rheum Dis. 2011 Sep;70(9):1613-8. doi: 10.1136/ard.2010.147694. Epub 2011 May 29. PMID 21623001